CLINICAL TRIAL: NCT06515899
Title: Association of Middle Molecules Clearance and Clinical Parameters With Haemodiafiltration Convection Volume
Brief Title: Association of Middle Molecules Clearance With HDF Volume
Status: Recruiting | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RD2023-68
Record Dates: First submitted 2024-02-16; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: End Stage Renal Disease
Keywords: Middle Molecules clearance in HDF; HDF; Middle molecules; beta 2 microglobulin; HDF convection volume
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HDF patients: ESRF patients who are receiving renal replacement therapy in the form of HDF

SUMMARY:
HDF is a dialysis technique which involves diffusion and convection. HDF with high convection volume has consistently shown to improve survival in dialysis patients in number of robust RCTs. The precise reason of this survival benefit remains unclear.

The investigators hypothesize that this survival benefit with high volume HDF is related to enhanced middle molecule clearance and hemodynamic stability. However, this relationship has not been studied so far.

This observational study is aimed to understand the relationship between HDF convection volume with middle molecules (Beta 2-Microglobulin) clearance during HDF.

Exploring the relationship of HDF volume with middle molecules clearance has significant clinical ramifications. Only a minority of patients are able to achieve target convection volume. Understanding these relationships can rationalize the HDF prescription from convection volume-based prescription to β2-Microglobulin clearance-based prescription which may be applicable to wider range of patients.

The relationship between pre-dialysis β2-Microglobulin levels and RKF offers the prospect of dispensing with pre- and post-dialysis urea and creatinine measurements and interdialytic urine collections, currently necessary for estimating RKF, thus simplifying its estimation.

β2-Microglobulin reduction ratio and its component pre and post-dialysis β2-Microglobulin levels could therefore provide a composite estimate of small and middle molecule clearance and RKF.

DETAILED DESCRIPTION:
People with severe kidney failure need treatment by dialysis or transplantation to stay alive. In the UK there are 25,000 people receiving treatment with haemodialysis (HD). Conventional haemodialysis works on the principle of diffusion for removal of toxins. Haemodiafiltration (HDF) is a technique of dialysis which implies the principle of convection in addition to diffusion. Large clinical trials comparing haemodiafiltration with conventional haemodialysis have reported better survival in patients having haemodiafiltration with large convection volume. The mechanism of survival benefit with high convection volume remains unclear.

The investigators hypothesize that the benefit of high convection volume haemodiafiltration is due to enhanced removal of large sized toxins called 'middle molecules'. Additionally, it may also be due to better blood pressure control and less inflammation when dialysing using this technique. The literature so far has been inconsistent to confirm this. Understanding the relationship of haemodiafiltration convection volume with middle molecules removal and clinical parameters is crucial for adoption of this mode of treatment. Additionally, it can potentially transform the presently imperfect dialysis prescription based on small molecule removal to clinically relevant middle molecules removal.

In this single centre cross sectional study, the investigators aim to recruit 400 adult participants who have been on haemodiafiltration for at least 3 months. Once consented, the participants will be observed in a single routine dialysis sessions (study visit) to record all the standard care clinical parameters and dialysis related information including dialysis convection volume from haemodiafiltration. Participants will also have routine blood tests at the start and end of the observed dialysis session and additional blood tests to measure the removal of middle molecules at the same time. The relationship of these observed clinical and measured toxins removal parameters with convection volume will be determined from the collected data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above.
* Ability to give informed consent.
* End stage renal failure treated by dialysis for at least 3 months.
* Established on hemodiafiltration for >4 weeks.
* Prognosis more than 6 months as assessed by PI

Exclusion Criteria:

* Age less than 18 years.
* Inability to give informed consent.
* Prognosis less than 6 months as assessed by PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End stage renal failure patient having renal replacement therapy in the form of Haemodiafiltration.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The relationship between HDF convection volume and β2 Microglobulin reduction ratio during a HDF session. | 18 months
The relationship between HDF convection volume and serum pre dialysis β2 Microglobulin concentration (measured in mg/L). | 18 months

SECONDARY OUTCOMES:
The relationship of HDF convection volume with average intradialytic blood pressure (mmHg). | 18 months
The relationship of HDF convection volume with average intradialytic core body temperature (degrees centigrade) | 18 months
The relationship of HDF convection volume with CRP (mg/L). | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Usama A Butt, MBBS, MRCP, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No